CLINICAL TRIAL: NCT02677792
Title: Wellness and Weight Family Group Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Principal Investigator, Crystal Stack Lim, Assistant Professor, University of Mississippi Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #2015-0155
Record Dates: First submitted 2016-02-02; First posted 2016-02-09 (Estimated); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Pediatric Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Behavioral Family Intervention (BFI) (Experimental)
  Interventions: Behavioral: Behavioral Family Intervention (BFI)

INTERVENTIONS:
Behavioral: Behavioral Family Intervention (BFI) — Participating families will receive standard medical care through the Wellness and Weight Clinic, as well as the BFI. The BFI is based on family systems (Minuchin et al., 1975) and social-cognitive (Bandura, 1998) theories. Each dyad will participate in simultaneous, but separate, 75-minute parent and child groups over a 3 month period. The groups will start off meeting every week for 8 weeks and then bi-weekly for 1 month. Thus, dyads will attend a total of 10 group meetings over the 3 month period (12.5 hours of total treatment contact).

SUMMARY:
The purpose of the current study is examine the feasibility and efficacy of providing a behavioral family intervention in 30 youth 10 to 17 years of age who are obese and attending a multidisciplinary pediatric obesity clinic and their parents. Participating families will complete assessments consisting of weight status, dietary intake, physical activity, health-related quality of life, psychological functioning, home-food environment, parenting skills, and self-efficacy at pre-treatment (Baseline), post-treatment (Month 3), and 2 month post-treatment follow-up (Month 5). Family attendance data will be collected during the behavioral family intervention and children and parents will complete a treatment satisfaction questionnaire at the post-treatment assessment. Health outcomes (e.g., A1C, glucose) routinely assessed through standard medical care in the multidisciplinary pediatric obesity clinic will be obtained from child medical charts.

ELIGIBILITY:
Inclusion Criteria:

1. child 10 to 17 years of age attending an outpatient pediatric obesity clinic visit
2. child or adolescent is obese (equal to or above the 95th percentile for BMI based on Centers for Disease Control and Prevention (CDC) norms for age and gender)
3. child or adolescent is accompanied by a parent or legal guardian
4. participating child and parent speak and read English
5. family agrees to attend group meetings at a medical clinic over a 3 month period

Exclusion Criteria:

1. participating child or parent, according to parent report, has dietary restriction or medical condition contraindicating mild energy restriction or moderate physical activity (e.g., musculoskeletal, heart, or respiratory condition, uncontrolled blood pressure or exercise induced asthma)
2. child diagnosed according to parent report with pervasive developmental delay (e.g., autistic disorder)
3. child or parent, according to parent report, in commercial weight loss program
4. child or parent currently prescribed medications to impact appetite or weight loss/gain, according to parent report
5. parent and child do not speak and read English

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2016-02; Primary Completion 2020-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Change in Child Weight Status (BMIz) | Baseline, Post-Treatment (Month 3), and Follow-up (Month 5)
  BMIz calculated from measured child height and weight

SECONDARY OUTCOMES:
Change in Total Child Physical Activity kcals from Block Kids Physical Activity Screener | Baseline, Post-Treatment (Month 3), and Follow-up (Month 5)
  Child-report questionnaire
Change in Child Dietary Intake Total kcals from 24-hour dietary recall | Baseline, Post-Treatment (Month 3), and Follow-up (Month 5)
  Child-report 24-hour dietary recall assessed via Automated Self-administered 24-hour recall (ASA24) System; Children will complete the ASA-2014-Kids
Change in Child A1C Values | Baseline, Post-Treatment (Month 3), and Follow-up (Month 5)
  From child medical chart - testing completed as part of standard medical care
Change in Child Glucose Values | Baseline, Post-Treatment (Month 3), and Follow-up (Month 5)
  From child medical chart - testing completed as part of standard medical care
Change in Parent Weight | Baseline, Post-Treatment (Month 3), and Follow-up (Month 5)
  Measured parent weight
Change in Total Parent Physical Activity kcals from Block Physical Activity Screener Adults | Baseline, Post-Treatment (Month 3), and Follow-up (Month 5)
  Parent-report questionnaire
Change in Parent Dietary Intake Total kcals from 24-hour dietary recall | Baseline, Post-Treatment (Month 3), and Follow-up (Month 5)
  Parent-report 24-hour dietary recall assessed via ASA24-2014

OTHER OUTCOMES:
Change in Child Self-Efficacy for Total Healthy Lifestyle Behaviors | Baseline, Post-Treatment (Month 3), and Follow-up (Month 5)
  Child-report questionnaire; sum of scores from Child Dietary Self-Efficacy Scale and Self-Efficacy for Physical Activity Scale
Change in Child-Reported Total Health-Related Quality of Life | Baseline, Post-Treatment (Month 3), and Follow-up (Month 5)
  Child-report; total score from Pediatric Quality of Life Inventory
Change in Parent-Reported Total Health-Related Quality of Life | Baseline, Post-Treatment (Month 3), and Follow-up (Month 5)
  Parent-report; total score from Pediatric Quality of Life Inventory
Change in Child Psychological Functioning (Total Problems Subscale from CBCL) | Baseline, Post-Treatment (Month 3), and Follow-up (Month 5)
  parent-report; Child Behavior Checklist (CBCL) Total Problems Scale
Change in Home Food Inventory Obesiogenic Food Availability Score | Baseline, Post-Treatment (Month 3), and Follow-up (Month 5)
  Parent-reported
Change in Total Parenting Competence | Baseline, Post-Treatment (Month 3), and Follow-up (Month 5)
  Parent-report; Total score from Parenting Sense of Competency (PSOC) Scale

CONTACTS AND LOCATIONS:
Overall Officials: Crystal S. Lim, Ph.D., Principal Investigator — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No